CLINICAL TRIAL: NCT06169761
Title: Assessment of Tongue Protrusion Motor Skills in Healthy Adult
Brief Title: Tongue Protrusion Assessment in Healthy Adult (FLEPI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, Principal Investigator, Université Catholique de Louvain
Other Study IDs: FLEPI
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Tongue; Motor skills; Protrusion; Strength; Fatigability
MeSH Terms: interventions — Risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults of 18 years and older will fill out the STOP-BANG Questionnaire and undergo protrusive motor skills measurements.
  Interventions: Other: Assessment of motor skills of the tongue and others muscles, see below) and risk for sleep apnea

INTERVENTIONS:
Other: Assessment of motor skills of the tongue and others muscles, see below) and risk for sleep apnea — The following items will be assessed:
  1. Risk for sleep apnea, through the STOP-BANG Questionnaire.
  2. Anthropometric data: Height, weight, neck circumference, maximal mouth opening and maximal mouth opening with tongue to palate (with the Quick Tongue-Tie Assessment tool).
  3. Tongue peak pressure (i.e., the maximal pressure - Pmax - exerted against the IOPI bulb in kPa) during 3 sec. of tongue protrusion and elevation.
  4. Tongue endurance (i.e., the time to task failure in maintaining a pressure equal to a fixed percentage of Pmax against the IOPI bulb) during tongue protrusion and elevation
  5. Tongue mobility restriction measured with the Quick Tongue-Tie Assessment Tool
  6. Maximum inspiratory and expiratory pressures measured with MicroRPM in cmH2O
  7. Handgrip strength (measured with a JAMAR dynamometer in kg)
  Tongue skills measurements will be repeated 2 to 4 weeks after baseline to assess the reliability of these measurements.

SUMMARY:
This study aims to evaluate tongue protrusion motor skills in healthy adults and to assess the reliability of these measurements as well as their validity in relation to other motor functions (handgrip and respiratory muscles).

DETAILED DESCRIPTION:
The tongue is an organ involved in multiple essential daily functions (such as eating, speaking, and breathing). Normative values exist for the motor skills of tongue elevation in individuals. However, data regarding protrusion are lacking. Yet, the protrusive strength of the tongue is of particular interest. Indeed a weak protrusive tongue strength may contribute to sleep apnea and swallowing disorders. Therefore, this study aims to collect normative and clinimetric (validity and reliability) data of tongue protrusion strength and endurance among healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older

Exclusion Criteria:

* Eating disorder
* Dysphagia
* Cardiorespiratory disorder
* Previous or ongoing obstructive sleep apnea-hypopnea syndrome
* Neurological conditions (including neuromuscular disorders)
* Previous or ongoing cancer of the head or neck
* Pregnancy
* Any physical or mental condition that may affect the ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprised healthy adults from Belgium, including both men and women aged 18 years and older, who meet all eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tongue protrusion peak pressure | Measured two times: at baseline and after 2 to 4 weeks
  Tongue peak pressure during protrusion movements will be measured via the IOPI device
Tongue protrusion endurance | Measured two times: at baseline and after 2 to 4 weeks
  Tongue endurance during protrusion movements will be measured via a timer (the time in seconds until the participant is not able to sustain tongue protrusion as controlled via the IOPI).

SECONDARY OUTCOMES:
Tongue elevation peak pressure | Measured two times: at baseline and after 2 to 4 weeks
  Tongue peak pressure during elevation movements will be measured via the IOPI device
Tongue elevation endurance | Measured two times: at baseline and after 2 to 4 weeks
  will be measured via a timer (the time in seconds until the participant is not able to sustain tongue protrusion as controlled via the IOPI).
Tongue mobility restriction | Measured once at baseline
  Assessed through the ratio between maximal mouth opening and maximal mouth opening with tongue to palate, measured with the Quick Tongue-Tie Assessment Tool
Maximum Inspiratory and Expiratory Pressure | Measured once at baseline
  Maximum Inspiratory and Expiratory pressure will be measured via the MicroRPM device
Handgrip Strength | Measured once at baseline
  Handgrip Strength will be measured with a JAMAR Hand Dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No